CLINICAL TRIAL: NCT01737788
Title: Randomised Trial of Cervical Cerclage With and Without Occlusion for the Prevention of Preterm Birth in Women Suspected for Cervical Insufficiency
Brief Title: Cervical Occlusion for the Prevention of Preterm Birth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to slow recruitment and an interim analysis showing no benefit of occlusion.
Sponsor: Niels Jørgen Secher (Other)
Responsible Party: Sponsor-Investigator, Niels Jørgen Secher, Professor, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CervOcc-001
Record Dates: First submitted 2012-11-24; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Uterine Cervical Incompetence
Keywords: Cervical cerclage; Uterine Cervical Incompetence
MeSH Terms: conditions — Uterine Cervical Incompetence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Trial (Experimental): Therapeutic cervical cerclage with or without cervical occlusion in women presenting with short cervix (<25mm)
  Interventions: Procedure: Cervical occlusion
- Prophylactic Trial (Experimental): Prophylactic cervical cerclage with or without cervical occlusion in women with a history of cervical insufficiency
  Interventions: Procedure: Cervical occlusion

INTERVENTIONS:
Procedure: Cervical occlusion — Women were randomized to receive cervical occlusion or no cervical occlusion in addition to a cervical cerclage (McDonald or Shirodkar cerclage). Cervical occlusion was performed with interrupted or continuous sutures, placed approximately 1 cm deep on each lip, and 0.5 cm apart with a nylon 2-0/3-0 suture.

SUMMARY:
The aim of this study was to evaluate the effect of cervical occlusion versus no cervical occlusion in women with cervical cerclages.

DETAILED DESCRIPTION:
Cervical weakness and ascending infection have long been considered important causes of preterm birth. Cervical occlusion could theoretically be used for the treatment of cervical weakness and to protect the cervix against infection. A cervical cerclage could be placed to increase the cervical resistance, and occlusion of the external os could be performed to retain the cervical mucus plug thereby preventing infection. The aim of this multicentre, stratified, randomised controlled trial was to evaluate the effect of cervical occlusion versus no cervical occlusion in women with prophylactic and therapeutic cervical cerclages.

ELIGIBILITY:
Inclusion Criteria:

* The physician in charge considered that a cerclage was indicated.
* Gestational age between 12 and 27 completed weeks.
* Previous late mid-trimester miscarriage, or spontaneous preterm labour and delivery before 28 weeks with or without previous cerclages.
* Previous cerclage because of short cervix.
* Confirmed gestational age defined as gestational age estimated by ultrasound at less than or equal to 22+0 weeks, and/or certain last menstrual period.
* Vaginal infection treated before cerclage.
* Ability to read and understand the relevant national language.
* Consent obtained in accordance with specifications of the local research ethics committee.
* 18 years or more of age and legally competent.

Exclusion Criteria:

* Demonstrated cervical infection.
* Obstetrical complications in the current pregnancy.
* Multiple pregnancies.
* History of a significant abruptio placenta in a previous pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2006-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Take-home baby rate | Neonates will be followed for the duration of stay in the neonatal intensive care unit, an expected average of 28 days with a minimum of 0 days up to a maximum of 98 days.
  Take-home baby rate was defined as the proportion of living babies discharged from the hospital of all singleton pregnancies.

SECONDARY OUTCOMES:
Gestational age at birth | At birth
  Evaluated as a continuous variable and as a dichotomous variable (<34+0 weeks gestation)

OTHER OUTCOMES:
Days of admission to the neonatal intensive care unit | Neonates will be followed for the duration of stay in the neonatal intensive care unit, an expected average of 28 days with a minimum of 0 days up to a maximum of 98 days.

CONTACTS AND LOCATIONS:
Overall Officials: Niels J Secher, Professor, Principal Investigator — Department of Obstetrics and Gynecology, Hvidovre University Hospital, Denmark
Locations (23):
- Adelaide, South Australia, Australia
- Denmark (14):
  - Odense, Funen
  - Aalborg, Jutland
  - Aarhus, Jutland
  - Horsens, Jutland
  - Kolding, Jutland
  - Viborg, Jutland
  - Copenhagen, Region Sjælland
  - Gentofte, Copenhagen, Region Sjælland
  - Glostrup, Copenhagen, Region Sjælland
  - Herlev, Copenhagen, Region Sjælland
  - Hillerød, Region Sjælland
  - Holbæk, Region Sjælland
  - Department of Obstetrics and Gynecology, Hvidovre University Hospital, Denmark, Hvidovre, Region Sjælland
  - Roskilde, Region Sjælland
- New Delhi, New Delhi, India
- Mecca, Mecca Region, Saudi Arabia
- Pretoria, Gauteng, South Africa
- Barcelona, Catalonia, Spain
- Malmo, Skåne County, Sweden
- Basel, Canton of Basel-City, Switzerland
- United Kingdom (2):
  - Liverpool, Lancashire
  - London, London

REFERENCES:
- [Derived] Brix N, Secher NJ, McCormack CD, Helmig RB, Hein M, Weber T, Mittal S, Kurdi W, Palacio M, Henriksen TB; CERVO group. Randomised trial of cervical cerclage, with and without occlusion, for the prevention of preterm birth in women suspected for cervical insufficiency. BJOG. 2013 Apr;120(5):613-20. doi: 10.1111/1471-0528.12119. Epub 2013 Jan 18. PMID 23331924